CLINICAL TRIAL: NCT01106885
Title: Effective Care Management of Depressed Diabetes Patients
Brief Title: Effective Care Management of Depressed Diabetes Patients (The Positive Steps Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency); Genesys Health System (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, John Piette, VA Senior Research Career Scientist and Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R18DK066166-01A1 (NIH); 1R18DK066166-01A1 (NIH)
Record Dates: First submitted 2010-04-15; First posted 2010-04-20 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Diabetes; Depression
Keywords: Diabetes; Depression; Telephone Care Management; Medication Care Management (MCM); Cognitive Behavioral Therapy (CBT)
MeSH Terms: conditions — Diabetes Mellitus; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced Usual Care (No Intervention): Adult patients with diabetes and depression.
  * Report screening results
  * Notify PCP of screening results (optional per patient)
  * PCP referrals
  * Educational materials regarding diabetes, physical activity, and depression
- Staged Care Management (Experimental): Adult patients with diabetes and depression
  Interventions: Behavioral: Medication Care Management (MCM); Behavioral: Cognitive-Behavioral Therapy (CBT)

INTERVENTIONS:
Behavioral: Medication Care Management (MCM) — * Basic physical activity counseling
  * Notify PCP and facilitate initiation of antidepressants
  * Medication monitoring calls at 1, 2, 4, 6, 8, 10, and 12 weeks*
  * 1/mo monitoring in continuation phase (mos. 4-12)*
  * Report & recommendations to PCP after each patient call
  * Note: *average of 10 minutes of telephone time each (series is repeated if second antidepressant trial is needed)
  Arms: Staged Care Management
Behavioral: Cognitive-Behavioral Therapy (CBT) — * Notify PCP
  * CBT Manual
  * Weekly CBT focused counseling for 12 weeks**
  * Monthly CBT in months 4-12**
  * Behavioral physical activity counseling
  * Report & recommendations to PCP after each patient call
  * Note: **average of 50 minutes of telephone time each
  Arms: Staged Care Management

SUMMARY:
Evaluation of telephone care management intervention designed to improve outcomes among depressed diabetes patients.

DETAILED DESCRIPTION:
Research Plan: 382 patients ages 21-80, including 177 women, and 123 Blacks from the Ann Arbor VA HCS, UM, and the Genesys Health Care System in Flint. Patients will be randomized to: (1) brief education about depression, diabetes self-care, and physical activity; or (2) telephone care management including antidepressant medication care management (MCM) and/or cognitive behavioral therapy (CBT). The MCM module uses a standard algorithm to identify efficacious antidepressants and promote adherence. The CBT module addresses symptoms, exercise, and communication skills.

Methods: Surveys: Patients will complete clinic-based surveys at baseline and 12-months to measure their health status, self-care, provider-patient communication, and resource use. At 4 months, they will complete a mailed questionnaire to capture short-term changes in depressive symptoms, walking, patient-provider communication, medication adherence, and quality-of-life. Physiologic Measures: At baseline and 12-months, patients' A1c and cholesterol will be measured via a fingerstick blood test. We also will measure blood pressure, height, and weight. With patients' 4-month mailed surveys, they will complete fingerstick A1c tests and return the results via mail. The blood tests are identical to those diabetes patients use to self-monitor their blood glucose. Pedometers: We will measure distance walked at baseline, 4 months, and 12 months using a pedometer. Patients will record their walk distances for one week and return the results via mail. Electronic data: Utilization and billing databases will be used to identify health service utilization (ER visits, outpatient care, hospitalizations) occurring during patients' participation and the prior 12 months. Physician feedback. At patients' 12-month assessment, the physician will complete a brief survey about the patient's communication style. All patients will provide written consent administered prior to their face-to-face screening and baseline interviews. Physician 12-month surveys about patients' communication style will be anonymous.

ELIGIBILITY:
Inclusion Criteria. Patients must meet all of the following criteria:

* Active Diabetes (Type 1 & 2)
* Diagnosis of depression
* Using hypoglycemic medications
* At least 1 outpatient visit in last 12 months
* At least 21 years old

Exclusion Criteria. Patients who have any of the following will be excluded:

* Limited life expectancy (heart failure/ on oxygen/ advanced stage cancer/ dialysis)
* End stage renal disease
* Lung cancer
* Dementia
* Bipolar
* Schizophrenia
* Can't speak English
* Memory problems
* Alcohol problems
* Illegal drug use
* Minimal depressive symptoms
* Blood pressure 180/110 or higher
* Problems with loss of consciousness
* Can't walk 10 minutes on level surface
* Not planning to get their care at study site
* PCP not affiliated with study site
* Are not on a stable regimen (change in depression Rx in last 28-30 days)
* Type 1 diabetic if diagnosed before age 15

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2005-05; Primary Completion 2009-10 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Participant HbA1c levels | one year
Participant cardiovascular risk index | one year

SECONDARY OUTCOMES:
Proximal intervention targets | one year
  (e.g., depressive symptoms, physical activity levels, and provider-patient communication)
Other self-care behaviors | one year
Health-related quality of life | one year
Treatment satisfaction | one year
Resource use | one year

CONTACTS AND LOCATIONS:
Overall Officials: John D Piette, PhD, Principal Investigator — VA Ann Arbor Healthcare System
Locations (3):
- United States (3):
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - University of Michigan Health System, Ann Arbor, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan

REFERENCES:
- [Derived] Piette JD, Valenstein M, Himle J, Duffy S, Torres T, Vogel M, Richardson C. Clinical complexity and the effectiveness of an intervention for depressed diabetes patients. Chronic Illn. 2011 Dec;7(4):267-78. doi: 10.1177/1742395311409259. Epub 2011 Aug 12. PMID 21840915